CLINICAL TRIAL: NCT04157413
Title: The Role of Essential Amino Acid Intake and Intestinal Permeability on Amino Acid Blood Profile and Linear Growth Among Indonesian Children 12-24 Months Living in an Agricultural Area: A Basis for a Food Based Intervention
Brief Title: Food-based Approach Development to Fulfil Amino Acid Gap by Considering the Intestinal Permeability of Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nia Novita Wirawan (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor-Investigator, Nia Novita Wirawan, Assistant Professor, University of Brawijaya
Organization: University of Brawijaya (Other)
Other Study IDs: l9-10-1169
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Stunting
Keywords: amino acid intake; blood amino acid; stunting; linear growth; intestinal permeability; lactulose mannitol ratio
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stunted Group: A comparative cross sectional study will compare stunted group and non-stunted group on amino acid intake, blood amino acid and intestinal permeability. Stunted group is defined as children who have LAZ <-2 SD
- Non-stunted Group: Non-stunted group will be those with LAZ >= 0.5 SD matching by age and sex with stunted group. Other criteria will be similar. No Intervention will be given to the groups in this proposed protocol.

SUMMARY:
This study will be comprised of 2 phases. Phase 1 study is a comparative cross-sectional study which will be conducted among children aged 12-24 months living in agricultural area. A total of 172 healthy children consisted of 86 stunted children (Length for age z-score <-2 Standard deviation) and 86 non-stunted children (Length for age z-score ≥0.5 Standard Deviation) will be recruited. Dietary intake, urine and dried blood spot from finger prick will be collected to assess amino acid intake, intestinal permeability and essential blood amino acid respectively. Qualitative study i.e. focus group discussion (FGD) and market survey will also be implemented. According to the result of phase 1 study, 2 types of food-based approaches will be developed, namely Complementary food recommendations (CFR) and Food multi-mix formula

DETAILED DESCRIPTION:
Phase 1 study will recruit a total of 172 healthy children who are matched by sex and age. Aside of being stunted, children must have normal weight for length z-score (not wasted or overweight). Data collection will be performed as follows:

1. Dietary intake of the children will be collected by 9 days Estimated Food Record by visiting the respondents house
2. Urine will be collected once to measure intestinal permeability profile using Lactulose Mannitol ratio indicator.
3. Dried blood spot from finger prick will be collected to essential blood amino acid.

To collect information on locally available and culturally accepted protein rich food sources, series of focus group discussion (FGD) and market survey will also be implemented.

Food-based approaches will be developed according to the information attained from phase 1 study. Problem nutrients that are identified from dietary assessment will be fulfilled through optimization of locally available food by using linear programming approach. Problem nutrients that are not able to be fulfilled by CFR will be use as a basis to develop a Food multi-mix (FMM) formula. Data of intestinal permeability profile will be used to add other locally available food in FMM that are potential to improve intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

1. Stunting group is defined as length for age Z-score (LAZ) <-2.0 SD and non-stunting group as LAZ ≥-0.5 SD
2. Normal weight for length Z-score (WLZ ≥-2 SD to ≤+1 SD)
3. Group matching by age, gender
4. Singleton
5. Full term gestation
6. Normal birth weight
7. Living with mother
8. Not suffered from diarrhea at least in the last 1 month (as reported by the mothers)
9. Not suffering from fever during assessment (as measured by the health staff)
10. Not born from diabetic mothers (as reported by the mothers)

Exclusion Criteria:

1. Drink Ultra High Temperature (UHT) milk at least 15 days before urine collection
2. Taking any medication.
3. Had taken non-steroidal anti-inflammatory drugs within two weeks of the study,
4. Taken antibiotics within 4 weeks of the study,
5. Unable to drink the sugar solution
6. Refuse to participate until completion of the study

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Target population of this study are children 12-24 months living in rural agricultural area in Kabupaten Malang. Kecamatan will be chosen based on the high prevalence of stunting and having potentials of protein food source to be optimized. Sample of the study are children living in selected villages in the period of 2019-2020 who fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2020-01-02 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Amino acid intake | January - February 2020
  Amino acid intake will be assessed by estimated food record
Blood amino acid | January - April 2020
  Essential blood amino acid will be measured from finger prick dried blood spot and will be analyzed using LC-MS/MS
Intestinal Permeability | January-April 2020
  Intestinal permeability will be measured from urine and will be analyzed using HPLC

OTHER OUTCOMES:
Linear growth | December 2019
  Linear growth in terms of length will be measured using anthropometric measurements to define stunted and non-stunted group.

CONTACTS AND LOCATIONS:
Overall Officials: Badriul S Hegar, Prof, Study Chair — Indonesia University

IPD SHARING:
Plan to Share IPD: No
I will not share the IPD of the subject participated due to consent issue